CLINICAL TRIAL: NCT05779124
Title: Soluble B-Cell Activating Factor and a Proliferation-inducing Ligand for Transplant Risk Assessment and Prediction of Antibody-Mediated Rejection in Kidney Transplantation: a Prospective Multicenter Cohort Study
Brief Title: BAFF/APRIL in Kidney Transplant Rejection Risk Assessment
Acronym: BA-TRAP
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The Shenzhen's People's Hospital (Unknown); Shenzhen Third People's Hospital (Other); Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Changxi Wang, Director of Department of Kidney Transplantation, Organ Transplant Center, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: sBA-KTX-2023
Record Dates: First submitted 2023-03-03; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplantation; Kidney Transplant Rejection
Keywords: kidney transplantation; soluble B lymphocyte activating factor; antibody-mediated rejection; a proliferation-inducing ligand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — We willl collect the peripheral blood samples from recipients for further biological research on the BAFF/APIRL pathway. The anonymized samples will be collected after obtaining informed consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antibody-mediated rejection (AMR) is a significant risk factor for graft loss in kidney transplantation. Soluble B cell-activating factor (sBAFF) and a proliferation-inducing ligand (APRIL) plays a critical role in the activation and differentiation of B cells, making it a potential predictive biomarker for AMR. In this prospective multicenter cohort study, the effectiveness of sBAFF/APRIL in predicting AMR after kidney transplantation is evaluated. Recipient sBAFF/APRIL levels are monitored before transplantation, and at seven days, two weeks, one month, three months, and every three months after transplantation continuously . The primary outcome is the occurrence of AMR, while the status of donor-specific antibodies (DSA), T cell-mediated rejection (TCMR), and other clinical parameters are secondary outcomes. The predictive capacity of sBAFF/APRIL for both the primary and secondary outcomes will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Living donor or deceased donor kidney recipients.
2. Patient is willing and capable of giving written informed consent for participation and able to participate in the study for 24 months.

Exclusion Criteria:

1. Preoperative donor specific antibody positive .
2. Combined or multi-organ transplantation.
3. Poor compliance.
4. Unable to continue the follow-up.
5. Patients who are judged by the doctors to be excluded for this trial (Details need to be provided).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplantation recipients
Sampling Method: Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Antibody-mediated Rejection | 24 months
  Antibody-mediated rejection is diagnosed based on kidney biopsy according to Banff 2019 criteria

SECONDARY OUTCOMES:
Incidence of de novo donor-specific antibody | 24 months
  Donor-specific antibody is monitored before transplantation and every six months after transplantation.
Incidence of T cell-mediated rejection | 24 months
  T cell-mediated rejection is diagnosed based on kidney biopsy according to Banff 2019 criteria
Incidence of infection | 24 months
Estimated glomerular filtration rate (eGFR) | 24 months
  eGFR is calculated based on Modification of Diet in Renal Disease (MDRD) formula, at one week, two weeks, one month, 3 months and every 3 months later, after kidney transplantation.
Qualitative or Quantitative meassurement of urine protein | 24 months
  Urine protein test result is collected at one week, two weeks, one month, 3 months and every 3 months later, after kidney transplantation.
Renal graft survival | 24 months
  Graft loss is defined as return to dialysis, removal of renal graft or kidney re-transplantation.
Death-censored renal graft survival | 24 months
  Death-censored renal graft survival is defined as graft survival censored for death with a functioning graft
Patient survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Changxi Wang, M.D., Ph.D., Study Chair — First affiliated hospital of Sun Yet-Sen university
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu S, Su X, Ye Q, Wei Y, Gao Y, Huang M, Chen Y, Wang J, Zhang Q, Fu Q, Li J, Wu C, Huang H, Xu B, Zhang H, Liu L, Wang C. Serum Soluble B Cell-Activating Factor Is a Non-Invasive Biomarker of Antibody-Mediated Rejection in Kidney Allograft With Satisfactory Risk Stratification Performance But Negligible Diagnostic Value. Front Immunol. 2022 Apr 13;13:869444. doi: 10.3389/fimmu.2022.869444. eCollection 2022. PMID 35493478
- [Background] Zhang H, Wang S, Su X, Fu Q, Li J, Wang J, Deng R, Wu C, Huang Q, Liu L, Wang C. The role of soluble B cell-activating factor in further stratifying the risk of antibody-mediated rejection post-renal transplant: A meta-analysis. Int Immunopharmacol. 2020 Feb;79:106059. doi: 10.1016/j.intimp.2019.106059. Epub 2019 Dec 20. PMID 31865240